CLINICAL TRIAL: NCT05081908
Title: Hypofractionated Stereotactic Radiotherapy (Multisession Radiosurgery) in Residual/Recurrent Grade II Meningiomas: Feasibility Study.
Brief Title: Multisession Radiosurgery in Residual/Recurrent Grade II Meningiomas.
Acronym: ATM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ATM
Record Dates: First submitted 2021-09-14; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Meningioma Atypical
Keywords: atypical meningioma; radiosurgery; multisession radiosurgery; recurrence meningioma
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multisession radiosurgery (Experimental): Radiosurgery
  Interventions: Procedure: Radiosurgery

INTERVENTIONS:
Procedure: Radiosurgery — Multisession radiosurgery (hypofractionated radiotherapy) with Cyberknife

SUMMARY:
Fractionated radiosurgery will be delivered to atypical meningioma lesions in salvage setting for patients who present post-surgical residual lesion or develop recurrence.

DETAILED DESCRIPTION:
Meningioma is the most common intracranial tumor (1). World Health Organization (WHO) grade II (atypical) meningioma recurs more frequently than WHO grade I (benign) meningioma, and patients with subtotally resected atypical meningioma should be treated with adjuvant radiation therapy (2). However, many atypical meningiomas can be gross totally resected, and whether to administer radiation to this population remains unclear. Apart from extent of resection, clinical characteristics such as age and gender and tumor-related characteristics such as tumor size and location have poor predictive capacity to determine which lesions will recur.

The lack of professional consensus on the role of adjuvant radiation therapy (RT) derived from the heterogeneity and retrospective nature of the published data: standard fractionation fails to demonstrate a benefit in term of local control and survival.

Recent advances in radiotherapy technology (staged radiosurgery) give the possibility to reach high dose levels only in tumor volume and in the same time to save the surrounding healthy tissues.

The purpose of this study is to verify the related toxicity of a new radiotherapy protocol and as second end point to evaluate the efficacy on disease local control at 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients had residual or recurrent atypical meningioma (grade II) after surgery (Simpson score)
* Age: ≥ 18 years old
* Karnofsky performance Status ( KPS) ≥ 70
* Written consent

Exclusion Criteria:

* Pregnancy
* Neurofibromatosis type 2 (NF2)
* Concomitant aggressive haematological or solid neoplasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-05-17 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Neurological side effects | through study completion, up to 2 year
  Frequency of neurological side effects related to the radiosurgical treatment, evaluated according with CTCAE scale at every follow-up (4 months post-treatment, then every 6 months).

SECONDARY OUTCOMES:
Local control | through study completion, up to 2 year
  The rate of tumor response defined as follow on the basis of modification of MRI imaging evaluated also with advanced RM techniques:Partial response (PR) is defined as 20%, decrease in the volumetric size of the lesion on MRI; stable disease (SD) as no change in the size of the lesion; progressive disease (PD) increase in any volumetric size of the lesion, confirmed at least a the following two consecutive MR

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Radioterapia, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ostrom QT, Gittleman H, Liao P, Rouse C, Chen Y, Dowling J, Wolinsky Y, Kruchko C, Barnholtz-Sloan J. CBTRUS statistical report: primary brain and central nervous system tumors diagnosed in the United States in 2007-2011. Neuro Oncol. 2014 Oct;16 Suppl 4(Suppl 4):iv1-63. doi: 10.1093/neuonc/nou223. No abstract available. PMID 25304271
- [Background] Aghi MK, Carter BS, Cosgrove GR, Ojemann RG, Amin-Hanjani S, Martuza RL, Curry WT Jr, Barker FG 2nd. Long-term recurrence rates of atypical meningiomas after gross total resection with or without postoperative adjuvant radiation. Neurosurgery. 2009 Jan;64(1):56-60; discussion 60. doi: 10.1227/01.NEU.0000330399.55586.63. PMID 19145156
- [Derived] Marchetti M, Pinzi V, Iezzoni C, Morlino S, Tramacere I, De Martin E, Cane I, Fariselli L. Multisession radiosurgery for grade 2 (WHO), high risk meningiomas. A phase II clinical trial. J Neurooncol. 2022 May;157(3):397-403. doi: 10.1007/s11060-022-03978-w. Epub 2022 Apr 4. PMID 35378640